CLINICAL TRIAL: NCT04555317
Title: Bone Toxicity Following Pelvic Radiotherapy: A Prospective Randomised Controlled Feasibility Study Evaluating a Musculoskeletal Health Package in Women With Gynaecological Cancers Undergoing Pelvic Radiotherapy
Brief Title: Bone Toxicity Following Pelvic Radiotherapy
Acronym: RadBone
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Christie NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CFTSp180
Record Dates: First submitted 2020-09-02; First posted 2020-09-18 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-08

CONDITIONS: Gynecologic Cancer; Radiotherapy Side Effect; Fracture
MeSH Terms: conditions — Radiation Injuries; Fractures, Bone

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned to either an observational arm or an interventional arm consisting of a musculoskeletal health package
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): No intervention. Standard of care cancer pathway followed.
- Musculoskeletal Health Package (Active Comparator): 3 month prehabilitation exercise program during radiotherapy and assessment of BMD at baseline with appropriate management according to fracture risk assessment (with either (a) lifestyle advice, (b) calcium and vitamin D (c) calcium, vitamin D and bisphosphonate (alendronate))
  Interventions: Combination Product: Musculoskeletal health package

INTERVENTIONS:
Combination Product: Musculoskeletal health package — 3 month prehabilitation exercise program during radiotherapy with assessment of BMD at baseline with appropriate management according to fracture risk assessment (with either (a) lifestyle advice, (b) calcium and vitamin D (c) calcium, vitamin D and bisphosphonate (alendronate))
  Arms: Musculoskeletal Health Package

SUMMARY:
A randomised controlled clinical feasibility trial to determine the feasibility and acceptability of a "musculoskeletal health package (MHP)" intervention in women undergoing pelvic radiotherapy for gynaecological malignancies and inform power calculations for a definitive trial.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years
* histologically confirmed uterine or cervix cancer
* patients undergoing potentially curative/adjuvant radiotherapy
* ability to give informed consent to participate

Exclusion Criteria:

* age less than 18 years or greater than 85 years
* patients with pre-existing bone conditions such as: osteoporosis treated with bisphosphonates in the previous 5 years/fibrous dysplasia/osteogenesis imperfecta or other metabolic bone condition
* inability to give informed consent to participate
* home address outside Greater Manchester
* contraindication or intolerance of Magnetic Resonance scanning

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Gynae-oncology patients with cervical or endometrial cancer
Enrollment: 80 (Estimated)
Dates: Start 2021-05-17 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Eligibility and screening rate | baseline
  proportion of patients eligible for the study from the patient population
Recruitment and study group allocation rate | 2 weeks post consent
  number of eligible patients recruited, randomised and allocated to appropriate study populations
Recruitment and study group allocation rate | 2 weeks post consent
  proportion of eligible patients recruited, randomised and allocated to appropriate study populations
Intervention fidelity rate | end of study 18 months
  number of patients completing the elements of the study
Intervention fidelity rate | end of study 18 months
  proportion of patients completing the elements of the study
Attrition rate | end of study 18 months
  number of patients lost to follow-up
Patient and physician acceptability y | change from baseline to 6 months
  Patient and physician acceptability assessed with electronic questionnaires
Patient and physician acceptability y | change from baseline to 12 months
  Patient and physician acceptability assessed with electronic questionnaires
Patient and physician acceptability y | change from baseline to 18 months
  Patient and physician acceptability assessed with electronic questionnaires
Health Economic QOL Analysis | change from baseline to 6 months
  EuroQol-5D-5L Quality of Life assessment
Health Economic QOL Analysis | change from baseline to 12 months
  EuroQol-5D-5L Quality of Life assessment
Health Economic QOL Analysis | change from baseline to 18 months
  EuroQol-5D-5L Quality of Life assessment

SECONDARY OUTCOMES:
Incidence of Radiotherapy Related Insufficiency Fracture (RRIF) | assessed at 6, 12 , 18 months post radiotherapy
  Incidence of RRIF assessed by MR
Longitudinal change in BMD | assessed at baseline and 18 months
  BMD measured by DXA at baseline and 18 months
Longitudinal change in fracture risk using FRAX (inc BMD by DXA) | assessed at baseline and 18 months
  FRAX assessment tool (including femoral neck BMD)
Longitudinal change in biochemical markers of bone turnover (BTM) | change from baseline to week 2
  serum Bone Turnover Markers
Longitudinal change in biochemical markers of bone turnover (BTM) | change from baseline to week 3
  serum Bone Turnover Markers
Longitudinal change in biochemical markers of bone turnover (BTM) | change from baseline to week 4
  serum Bone Turnover Markers
Longitudinal change in biochemical markers of bone turnover (BTM) | change from baseline to week 5
  serum Bone Turnover Markers
Longitudinal change in biochemical markers of bone turnover (BTM) | change from baseline to week 6
  serum Bone Turnover Markers
Longitudinal change in biochemical markers of bone turnover (BTM) | change from baseline to week 7
  serum Bone Turnover Markers
Longitudinal change in biochemical markers of bone turnover (BTM) | change from baseline to week 8
  serum Bone Turnover Markers
Longitudinal change in biochemical markers of bone turnover (BTM) | change from baseline to week 9
  serum Bone Turnover Markers
Longitudinal change in biochemical markers of bone turnover (BTM) | change from baseline to 6 months
  serum Bone Turnover Markers
Longitudinal change in biochemical markers of bone turnover (BTM) | change from baseline to 12 months
  serum Bone Turnover Markers
Longitudinal change in biochemical markers of bone turnover (BTM) | change from baseline to 18 months
  serum Bone Turnover Markers
Quality of Life Assessment : adapted CTCAE pelvic questionnaire | change from baseline to 6 months
  CTCAE pelvic questionnaire, (common terminology criteria for adverse events). (measures: Bowel questions scored out of 22, urinary questions out of 19 and sexual questions out of 8. Total out of 49: higher score = worse quality of life)
Quality of Life Assessment : adapted CTCAE pelvic questionnaire | change from baseline to 12 months
  CTCAE pelvic questionnaire, (common terminology criteria for adverse events). (measures: Bowel questions scored out of 22, urinary questions out of 19 and sexual questions out of 8. Total out of 49: higher score = worse quality of life)
Quality of Life Assessment : adapted CTCAE pelvic questionnaire | change from baseline to 18 months
  CTCAE pelvic questionnaire, (common terminology criteria for adverse events). (measures: Bowel questions scored out of 22, urinary questions out of 19 and sexual questions out of 8. Total out of 49: higher score = worse quality of life)
Quality of Life Assessment: SMFA adapted to lower limbs | change from baseline to 6 months
  adapted SMFA : short form musculoskeletal function assessment (scores are standardised with high scores indicating poor function. 39 questions min score possible 39, max score possible 195 (raw scores)
Quality of Life Assessment: SMFA adapted to lower limbs | change from baseline to 12 months
  adapted SMFA : short form musculoskeletal function assessment (scores are standardised with high scores indicating poor function. 39 questions min score possible 39, max score possible 195 (raw scores)
Quality of Life Assessment: SMFA adapted to lower limbs | change from baseline to 18 months
  adapted SMFA : short form musculoskeletal function assessment (scores are standardised with high scores indicating poor function. 39 questions min score possible 39, max score possible 195 (raw scores)

CONTACTS AND LOCATIONS:
Locations (1):
- Christie Hospital NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification will be available, according to below sponsor requirements: onsent to share data from this study for future research is voluntary. To ensure compliance with regulatory and governance requirements, approval from the sponsor team is required prior to the release of any data generated by this Christie sponsored study, to a third party. Any requests are to be directed towards the-christie.sponsoredresearch@nhs.net for consideration and must follow all local Policies and review procedures. If a proposal is accepted, then the sponsor will work with the requestor to develop any necessary data transfer plans/agreements.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will become available following analysis and initial publication of study findings. No end date.
Access Criteria: Consent to share data from this study for future research is voluntary. To ensure compliance with regulatory and governance requirements, approval from the sponsor team is required prior to the release of any data generated by this Christie sponsored study, to a third party. Any requests are to be directed towards the-christie.sponsoredresearch@nhs.net for consideration and must follow all local Policies and review procedures. If a proposal is accepted, then the sponsor will work with the requestor to develop any necessary data transfer plans/agreements.

REFERENCES:
- [Derived] Chatzimavridou Grigoriadou V, Barraclough LH, Baricevic-Jones I, Bristow RG, Eden M, Haslett K, Johnson K, Kochhar R, Merchant Z, Moore J, O'Connell S, Taylor S, Westwood T, Whetton AD, Yorke J, Higham CE. RadBone: bone toxicity following pelvic radiotherapy - a prospective randomised controlled feasibility study evaluating a musculoskeletal health package in women with gynaecological cancers undergoing pelvic radiotherapy. BMJ Open. 2022 Jun 14;12(6):e056600. doi: 10.1136/bmjopen-2021-056600. PMID 35701060